CLINICAL TRIAL: NCT03394469
Title: Sarcopenic Obesity: Estimation of Prevalence and Identification of Clinical and Biological Determinants in a Population of Adult Obese Patients
Acronym: OBESAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHU-366; 2017-A01510-53. (Other: 2017-A01510-53.)
Record Dates: First submitted 2017-11-16; First posted 2018-01-09 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Obesity; Sarcopenia
MeSH Terms: conditions — Obesity; Sarcopenia

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort (Other): Collection of clinical and paraclinical data (biological and anthropometric) for evaluation of sarcopenic obesity in obese patients.
  Interventions: Other: collection

INTERVENTIONS:
Other: collection — Blood, urinary and faecal samples

SUMMARY:
This project aims first to determine the prevalence of sarcopenia in a population of obese people of extended age group (18-70 years). In a second step, the factors determining and / or predisposing to sarcopenic obesity will be identified as well as plasmatic and urinary biomarkers specific to this phenotype.

DETAILED DESCRIPTION:
Collection of clinical and paraclinical data (biological and anthropometric) for evaluation of sarcopenic obesity in obese patients.

Biological collection to identify plasma, serum, genetic, urinary and faecal biomarkers associated with sarcopenic obesity

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Sex: men and women
* Patient followed in clinical nutrition benefiting from a metabolic assessment for optimization of clinical and paraclinical management
* Patient meeting the criteria of obesity defined by BMI> 30 kg / m²
* Major patient with free, informed and signed consent
* Patient covered by the social security scheme

Exclusion Criteria:

* Patient with cancer or severe chronic disease (renal failure, respiratory failure, liver failure)
* Patient with neuromuscular disease
* Patient with a total inability to walk
* Minor patient
* Refusal of the patient to participate in the study
* Pregnant or lactating women
* Patient deprived of liberty or under guardianship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-06-06 (Estimated); Study Completion 2020-06-06 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia | at day 1
  The primary endpoint is sarcopenia (present / absent), defined using the muscle mass index (SMI) corresponding to = SM / Height², where the total muscle mass (SM) is calculated from validated equations. by Janssen et al in a population of men and women with a large age range (18-86 years) and adiposity (BMI: 16-48 kg / m integrating bio-impedancemetry data ( BIA).

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France